CLINICAL TRIAL: NCT01352741
Title: Evaluation of the Effectiveness, Safety, and Tolerability of Tapentadol PR Versus a Combination of Tapentadol PR and Pregabalin in Subjects With Severe Chronic Low Back Pain With a Neuropathic Pain Component
Brief Title: Comparison of Increasing Doses of Tapentadol Versus a Combination of Tapentadol and Pregabalin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 247251; 2010-019998-14 (EudraCT Number); KF5503/58 (Other: Grünenthal GmbH)
Record Dates: First submitted 2011-04-12; First posted 2011-05-12 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain; Neuropathic Pain
Keywords: low back pain; neuropathic; pain assessment; centrally acting tapentadol pregabalin; severe chronic
MeSH Terms: conditions — Low Back Pain; Neuralgia; Bronchiolitis Obliterans Syndrome | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tapentadol Prolonged Release (Experimental): Tapentadol Prolonged Release (100 - 500 mg per day) Oral administration twice daily
  Interventions: Drug: Tapentadol Prolonged Release; Drug: Tapentadol Prolonged Release open label maintenance
- Tapentadol Prolonged Release with Pregabalin (Active Comparator): Tapentadol Prolonged Release (100 - 300 mg per day) with Pregabalin (150 - 300 mg per day) Both administered orally twice a day.
  Interventions: Drug: Tapentadol Prolonged Release with Pregabalin; Drug: Tapentadol Prolonged Release open label maintenance

INTERVENTIONS:
Drug: Tapentadol Prolonged Release — 100 - 500 mg per day orally twice daily for a maximum of 12 weeks
  Arms: Tapentadol Prolonged Release
Drug: Tapentadol Prolonged Release with Pregabalin — Tapentadol Prolonged Release 100 - 300 mg per day with Pregabalin 150 - 300 mg per day orally twice daily for a maximum of 12 weeks
  Arms: Tapentadol Prolonged Release with Pregabalin
Drug: Tapentadol Prolonged Release open label maintenance — 100 - 400 mg per day Tapentadol Prolonged Release orally administered twice daily

SUMMARY:
The main objective of the study is to evaluate the effectiveness, safety, and tolerability of increasing doses of tapentadol prolonged release (PR) (500 mg per day) versus a combination of tapentadol PR (300 mg per day) and pregabalin (to 300 mg per day) in subjects requiring additional analgesia after titration to tapentadol PR 300 mg per day.

This is a clinical effectiveness trial designed to establish a link between anticipated clinical outcomes and the clinical practice by means of selected measures of clinical and subject reported outcomes. Since, severe low back pain with a neuropathic component, the targeted study population, is frequently treated with a combination therapy (monotherapy is often not effective enough) it is of interest to determine if tapentadol alone (combining 2 mechanisms of action in a single molecule) could be as effective as a combination of tapentadol plus pregabalin. Furthermore, the tolerability profiles of monotherapy versus combination are of interest.

DETAILED DESCRIPTION:
Participants with a diagnosis of chronic low back pain (defined as pain lasting for at least 3 month) and requiring a strong analgesic (World Health Organization [WHO] Step III) as judged by the investigator and having a positive or unclear score using the painDETECT diagnostic screening questionnaire will enter the open-label titration tapentadol prolonged release (PR) period. In total participants will have 11 planned scheduled visits scheduled over 105 days. At the Enrollment Visit [Day -14 (3 to 14 days prior to the Baseline Visit)] the inclusion and exclusion criteria will be checked to evaluate the participant's eligibility for the trial. Participants on previous analgesics will start a washout period three days up to 2 weeks.The duration of the washout period will depend on previous opioid analgesics and co-analgesics and their respective doses, down-tapering steps. Participants who do not need a washout of previous analgesic treatment (e.g. WHO Step I analgesics), a baseline visit can be scheduled as soon as clinical laboratory monitoring results are available.

At the Baseline Visit (Day 1) participants will start the 3 week open-label titration period tapentadol prolonged release (PR) at doses of 2 x 50 mg per day and will be titrated upwards in steps of 100 mg (2 x 50 mg) on a weekly basis.

Participants who do not qualify for randomization may continue the trial in the open-label continuation arm if they have already reached a satisfactory level of pain relief.

Participants qualifying for randomization in the comparative period (Day 22 to 77) will be allocated to 1 of 2 treatment arms and will continue treatment.

Either they continue on tapentadol prolonged release (PR) with increasing doses of tapentadol PR

* After the randomization visit, participants will titrate up to a total daily dose of 400 mg.
* 1 week after the randomization visit, will titrate up to a total daily dose of 500 mg. Participants in this treatment arm will receive a final dose of 500 mg tapentadol PR per day.

Or start on a combination of tapentadol PR 300 mg per day with pregabalin

* After the randomization visit, participants will continue their previous regimen of tapentadol PR 2 x 150 mg per day plus pregabalin 2 x 75 mg (total daily dose of 150 mg pregabalin).
* 1 week after the randomization visit, participants will continue their previous regimen (end of titration period) of tapentadol PR 2 x 150 mg per day plus pregabalin 2 x 150 mg (total daily dose of 300 mg pregabalin). Participants in this treatment arm will receive a final dose of 300 mg tapentadol PR and 300 mg pregabalin.

Participants in the Comparative Period can be assigned to the open-label pick-up arm and will be treated with a stable dose of tapentadol PR 300 mg per day or 400 mg per day if they experience treatment emergent adverse events (at least possibly related to investigational medicinal product).The open-label pick-up period theoretically starts on Day 29, i.e. one week after the Randomization Visit.

The Final Evaluation (Day 77) is planned to take place 8 weeks after randomization.

After the Final Evaluation a Follow-up Period (blinded tapering down/out of IMP in Week 12 and Follow-up Visit (up to Day 91) will take place. Tapering down/out of medication will be performed according to the Summary of Product Characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of chronic low back pain; chronic pain defined as pain lasting for at least 3 months.
* Subject's pain must require a strong analgesic (defined as World Health Organization (WHO) step III) as judged by the investigator.
* The painDETECT diagnostic screening questionnaire score must be:

  * "positive" or
  * "unclear".or If the subject is being treated with a stable regimen of centrally acting analgesics (opioids) and/or co-analgesics, even a "negative" painDETECT score (but of at least 9) at the enrollment visit will be acceptable.
* If under regular daily pretreatment with a WHO step II/step III opioid analgesic and/or a centrally acting co-analgesic:

  * Subjects must be taking a WHO step II or step III analgesic or co- analgesic on a daily basis for at least 2 weeks prior to the enrollment visit.
  * Subjects pretreated with a WHO step II opioid analgesic and/or a centrally acting co-analgesic must have reported an average pain intensity score of at least 5 points (NRS-3≥5) during the last 3 days prior to the enrollment visit. or If under regular, daily pretreatment with a WHO step I analgesic monotherapy or if no regular analgesic pretreatment is reported:
  * Subjects must have an average pain intensity score of at least 6 points NRS-3≥6) in the last 3 days prior to the enrollment visit.

Exclusion Criteria:

* Presence of concomitant painful conditions other than low back pain that could confound the subject's trial assessments or self-evaluation of the index pain, e.g., syndromes with widespread pain such as fibromyalgia.
* Low back pain caused by cancer and/or metastatic diseases.
* Any painful procedures planned during the trial period (e.g., major surgery) that may, in the opinion of the investigator, affect the effectiveness or safety assessments of the Investigational Medicinal Product (IMP).
* Pending litigation or application for insurance/governmental benefits due to chronic pain or disability and, if granted, benefits might be influenced by a successful participation in the trial.
* Rare hereditary problems of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption, lactose intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Baron, Prof. Dr., Principal Investigator — Neurological pain research and therapy Clinic for Neurology Campus Kiel, University Clinic Schleswig-Holstein, Schittenhelmstr. 10, 24105 Kiel, Germany
Locations (59):
- Austria (6):
  - Site 506, Klagenfurt
  - Site 503, Senftenberg
  - Site 501, Vienna
  - Site 502, Vienna
  - Site 504, Vienna
  - Site 505, Vienna
- Belgium (5):
  - Site 605, Dour
  - Site 602, Genk
  - Site 603, Gozée
  - Site 604, Ham
  - Site 601, Pellenberg
- Denmark (4):
  - Site 702, Copenhagen
  - Site 704, Frederiksberg
  - Site 701, Glostrup Municipality
  - Site 703, Ringsted
- Germany (17):
  - DE 118, Berlin
  - Site 107, Berlin
  - Site 111, Böhlen
  - Site 105, Cologne
  - Site 116, Cologne
  - Site 115, Cottbus
  - Site 103, Hamburg
  - Site 110, Hamburg
  - Site 101, Kiel
  - Site 114, Kiel
  - Site 113, Leipzig
  - Site 109, Lübeck
  - Site 106, Rendsburg
  - Site 108, Schönau
  - Site 117, Weimar
  - Site 112, Westerstede
  - Site 104, Wiesbaden
- Netherlands (5):
  - Site 803, Amsterdam
  - Site 804, Eindhoven
  - Site 805, Enschede
  - Site 802, Heerenveen
  - Site 801, Sliedrecht
- Poland (12):
  - Site 309, Bydgoszcz
  - Site 312, Gdansk
  - Site 303, Katowice
  - Site 308, Krakow
  - Site 310, Krakow
  - Site 311, Krakow
  - Site 307, Lublin
  - Site 306, Ostrów Mazowiecka
  - Site 304, Poznan
  - Site 301, Warsaw
  - Site 302, Warsaw
  - Site 305, Wroclaw
- Spain (10):
  - Site 904, A Coruña
  - Site 908, Alicante
  - Site 901, Badalona
  - Site 905, Barcelona
  - Site 902, Centelles
  - Site 907, Granada
  - Site 909, Madrid
  - Site 910, Madrid
  - Site 903, Oviedo
  - Site 911, Valencia

REFERENCES:
- [Result] Baron R, Martin-Mola E, Muller M, Dubois C, Falke D, Steigerwald I. Effectiveness and Safety of Tapentadol Prolonged Release (PR) Versus a Combination of Tapentadol PR and Pregabalin for the Management of Severe, Chronic Low Back Pain With a Neuropathic Component: A Randomized, Double-blind, Phase 3b Study. Pain Pract. 2015 Jun;15(5):455-70. doi: 10.1111/papr.12200. Epub 2014 Apr 17. PMID 24738609
- [Result] Baron R, Kern U, Muller M, Dubois C, Falke D, Steigerwald I. Effectiveness and Tolerability of a Moderate Dose of Tapentadol Prolonged Release for Managing Severe, Chronic Low Back Pain with a Neuropathic Component: An Open-label Continuation Arm of a Randomized Phase 3b Study. Pain Pract. 2015 Jun;15(5):471-86. doi: 10.1111/papr.12199. Epub 2014 Apr 18. PMID 24750558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 23 Mar 2011 and the last participant completed the last follow-up examination on the 17 Jan 2012.
Pre-assignment Details: 622 participants signed an informed consent. All participants included in the 8 week Double Blind Comparative Period were initially in the open-label titration period.
  Participants in the open-label tapentadol continuation period were in the open-label titration period but did not enter the comparative period.
Groups:
- Tapentadol Prolonged Release: All participants entered the 3-week Titration Period, Tapentadol Prolonged Release was administered in an open-label fashion. Participants that did not qualify for entry into the Comparative Period were able to enter the open-label Continuation Period. During the double-blind comparator phase the dose was increased to 200 mg twice daily and after a week to 250 mg twice daily. Participants that dropped out due to tolerability issues during the comparative period were able to enter the open-label pick-up arm.
- Tapentadol Prolonged Release and Pregabalin: At the end of the Open-label Tapentadol Titration Period participants that qualified were randomized to either tapentadol or tapentadol and pregabalin treatment. In this double-blind period participants started on Tapentadol Prolonged Release 300 mg per day (2 x 150 mg) plus Pregabalin 2 x 75 mg (total daily dose of 150 mg). A week later the dose of Pregabalin was increased to a total daily dose of 300 mg per day (2 x 150 mg), the Tapentadol Prolonged Release dose remained at 300 mg per day.
Period: Open-label Tapentadol Titration Period
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Started | 445 (All participants started with 2 x 50 mg tapentadol PR and titrated upwards in steps of 100 mg/day.) | 0
Switched to Open-label Continuation Arm | 59 | 0
Full Analysis Set | 436 | 0
Completed | 372 (59 of 73 participants not completing the titration period entered the open-label continuation arm.) | 0
Not Completed | 73 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Lack of Efficacy | 19 | 0
Not completed — Adverse Event | 34 | 0
Not completed — Withdrawal of consent | 7 | 0
Not completed — Non-compliance with Trial Requirements | 5 | 0
Not completed — Other | 4 | 0
Period: Double-blind Comparative Period
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Started | 154 (Of the 313 participants that qualified for randomization 154 were randomized to tapentadol.) | 159 (159 of the 313 participants that qualified were randomized to tapentadol and pregabalin treatment.)
Switched to Open-label Pick-up Arm | 19 | 18
No Pain Assessments Available | 2 | 2
Full Analysis Set | 152 | 157
Major Protocol Deviations | 13 | 8
Per Protocol Set | 139 | 149
painDetect Per Protocol Set | 109 | 127
SF-12 Per Protocol Set | 131 | 143
EQ-5D Per Protocol Set | 131 | 143
HADS Per Protocol Set (PPS) | 123 | 137
Sleep Evaluation (Latency) PPS | 123 | 137
Sleep Evaluations (Awakenings) PPS | 123 | 137
Sleep Evaluations (Hours Slept) PPS | 123 | 137
Completed | 126 | 133
Not Completed | 28 | 26
Not completed — Protocol Violation | 2 | 0
Not completed — Lack of Efficacy | 0 | 3
Not completed — Adverse Event | 16 | 17
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal of consent | 8 | 3
Not completed — Other | 1 | 2
Period: Open-Label Tapentadol Continuation Arm
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Started | 59 (59 of the 73 participants that did not qualify for the comparative period entered this arm.) | 0 (In this period no tapentadol PR and pregabalin treatment was planned by the protocol.)
Major Protocol Deviation | 2 | 0
Full Analysis Set | 57 | 0
Completed | 51 | 0
Not Completed | 8 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 0
Period: Open-Label Tapentadol Pick-Up Arm
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Started | 37 (19 from tapentadol in the comparative phase and 18 from tapentadol & pregabalin entered this arm.) | 0 (Participants did not continue treatment. They were switched to tapentadol PR or discontinued.)
Completed | 37 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Trial Participants: All participants that received at least one dose of tapentadol prolonged release at baseline, in the open-label titration period.
Arm/Group | All Trial Participants
Number analyzed (Participants) | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262
  Male | 183
Race/Ethnicity, Customized [Number; unit: participants]
  White | 441
  Asian | 2
  Other | 2
Region of Enrollment [Number; unit: participants]
  Spain | 54
  Belgium | 45
  Poland | 102
  Denmark | 41
  Austria | 55
  Netherlands | 26
  Germany | 122
Height [Mean (Standard Deviation); unit: cm] — Data available for 441 participants
  cm | 168.2 (9.97)
Weight [Mean (Standard Deviation); unit: kg] | 83.61 (17.542)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Data available for 441 participants.
  kg/m² | 29.57 (5.616)
Diagnosis of Lumbar Radiculopathy [Number; unit: participants] — Number of participants with dermatomal pain present as assessed by the investigator. For a participant to have diagnosed lumbar radiculopathy pain, they must have answered 'yes' to all three dermatomal pain questions and 'yes' to at least one of the three root dysfunction questions
  participants
    Yes | 310
    No | 134
    Missing | 1
History of low back pain [Median (Full Range); unit: years] — Participants were asked since when they suffer from their current pain.
  years | 6.3 [2.1 to 11.7]
Subject's satisfaction with previous treatment [Number; unit: participants]
  Poor | 126
  Fair | 233
  Good | 68
  Very Good | 10
  Excellent | 1
  Missing | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in the Average Pain Intensity Score for the Overall Low Back Pain on an 11-point Numeric Rating Scale (NRS-3)
Description: The primary endpoint is defined as the comparison of tapentadol prolonged release (PR) 300 mg plus 200 mg per day and the combination of tapentadol PR 300 mg per day and pregabalin 300 mg per day regarding the change in NRS-3 pain intensity scores (recalled average pain intensity score during the last 3 days on 11-point NRS, where 0 is the no pain and 10 is pain as bad as you can imagine) from the randomization visit to the final evaluation visit.
  Theoretically a maximum decrease of -10 and an increase of +4 in the pain intensity would have been possible. A negative sign indicates a decrease in pain intensity from the start of treatment. The higher the absolute values, the greater the change since the start of treatment (Baseline visit).
Time Frame: Randomization (Day 22); Final Evaluation Visit (Day 77)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol Prolonged Release: Tapentadol PR (100 - 300 mg per day) oral administration twice daily in the open-label titration period. Subsequently increased in the comparative period to Tapentadol Prolonged Release to 500 mg per day.
- Tapentadol Prolonged Release and Pregabalin: Tapentadol Prolonged Release (100 - 300 mg per day) in the open-label titration period. Subsequently Tapentadol 300 mg per day was combined with Pregabalin at a daily dose of 300 mg per day.
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale | -1.6 (2.52) | -1.7 (2.48)

2. Secondary Outcome: Open-label Titration Period: Average Pain Intensity Score for the Overall Low Back Pain on an 11-point Numeric Rating Scale (NRS-3)
Description: The recalled average pain intensity score on the NRS-3 was assessed using an 11-point Numeric Rating Scale (NRS). This scale recalls the average pain intensity during the last 3 days. The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your pain on average during the last 3 days (the last 72 hours prior to the visit)". Where 0 = no pain and 10 indicates pain as bad as you can imagine. This is the treatment period prior to the primary outcome period.
Time Frame: Enrollment (Day -14); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed values.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol Prolonged Release: Tapentadol PR (100 - 300 mg per day) oral administration twice daily. Tapentadol PR was administered in an open-label fashion during the 3-week titration period. All participants started at 2 x 50 mg (100 mg per day) after the baseline visit and titrated upwards on a weekly basis by 2 x 50 mg. Dose adjustment could have taken place after 3 days on a stable dose if the participant's pain required faster titration.
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 445
units on a scale
  Enrollment Visit (N=438) | 7.2 (1.21)
  Baseline Visit (N=440) | 8.3 (1.14)
  Randomization Visit (N=377) | 5.4 (1.83)

3. Secondary Outcome: Open-label Continuation Period: Average Pain Intensity Score for the Overall Low Back Pain on an 11-point Numeric Rating Scale (NRS-3)
Description: The recalled average pain intensity score on the NRS-3 was assessed using an 11-point Numeric Rating Scale (NRS). This scale recalls the average pain intensity during the last 3 days. The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your pain on average during the last 3 days (the last 72 hours prior to the visit)". Where 0 = no pain and 10 indicates pain as bad as you can imagine.
Time Frame: Enrollment (Day -14); Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Observed values.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol Prolonged Release: Participants that did not qualify for randomization to the Comparator Period, continued on a stable dose of Tapentadol Prolonged Release 300 mg per day, if they had reached a satisfactory level of pain relief.
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 59
units on a scale
  Enrollment Visit (N=56) | 7.3 (1.30)
  Baseline Visit (N=57) | 7.9 (1.23)
  Randomization Visit (N=57) | 2.6 (1.27)
  Final Evaluation Visit (N=59) | 2.6 (2.09)

4. Secondary Outcome: End of Open-label Pick-up Period: Average Pain Intensity Score for the Overall Low Back Pain on an 11-point Numeric Rating Scale (NRS-3)
Description: as for outcome 3
Time Frame: Final Evaluation Visit (Day 77)
Population: Observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol Prolonged Release After Tapentadol: Participants that drop-out of the double-blind tapentadol prolonged release treatment in the Comparative Period, due to tolerability issues, continued on Tapentadol Prolonged Release at either 300 mg per day or 400 mg per day in this Open-Label Pick-up arm.
- Tapentadol Prolonged Release After Tapentadol and Pregabalin: Participants that dropped-out of the Tapentadol Prolonged Release and Pregabalin in the double-blind Comparative Period continued with Tapentadol Prolonged Release at either 300 or 400 mg per day in this Open-Label Pick-up arm.
Arm/Group | Tapentadol Prolonged Release After Tapentadol | Tapentadol Prolonged Release After Tapentadol and Pregabalin
Number analyzed (Participants) | 19 | 18
units on a scale | 4.4 (2.83) | 4.5 (1.96)

5. Secondary Outcome: Open-label Titration Period: Radiating Pain
Description: The NRS-3 pain intensity score at the visits in the open-label titration period for the two comparative double-blind period treatment groups analyzed is reported. NRS-3 pain intensity score (recalled average pain intensity score during the last 3 days on an 11-point NRS) for radiating pain (pain radiating into or towards the leg, typically of shooting, radiating character, usually radiating below the knee towards the foot) is reported. Where 0 = no pain and 10 indicates pain as bad as you can imagine.
Time Frame: Enrollment Visit (Day -14); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 445
units on a scale
  Enrollment Visit (N=438) | 7.0 (1.64)
  Baseline Visit (N=440) | 8.0 (1.60)
  Randomization Visit (N=377) | 5.3 (2.16)

6. Secondary Outcome: Open-label Titration Period: Radiating Mean Pain Intensity Score for the Comparative Period Population
Description: as for outcome 5
Time Frame: Enrollment Visit (Day -14); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 7.1 (1.75) | 6.9 (1.49)
  Baseline Visit (N=139; N=149) | 8.1 (1.84) | 8.1 (1.37)
  Randomization Visit (N=139; N=149) | 5.6 (1.87) | 5.7 (1.86)

7. Secondary Outcome: Double-blind Comparative Period: Change in NRS-3 Pain Intensity Score for the Radiating Pain
Description: NRS-3 pain intensity score (recalled average pain intensity score during the last 3 days on 11-point NRS, where 0 is the no pain and 10 is pain as bad as you can imagine) for radiating pain (pain radiating into or towards the leg, typically of shooting, radiating character, usually radiating below the knee towards the foot).
  The value reported represents the change from the randomization visit (i.e., the last 3 days in the titration period) to the end of the double-blind comparative period (i.e., the last 3 days in the comparative period). The theoretical values range from -10 to 10. A negative sign indicates a decrease in pain from the start of treatment. The higher the absolute values, the greater the change since the start of treatment (baseline visit).
Time Frame: Randomization Visit (Day 22); End of Evaluation Visit (Day 77)
Population: Double-blind comparative population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale | -1.5 (2.61) | -1.9 (2.60)

8. Secondary Outcome: Open-label Titration Period: Worst Mean Pain Intensity Scores Over the Past 24 Hours
Description: The recalled worst pain intensity during the last 24 hours was assessed using an 11-point Numeric rating scale, where 0 = no pain and 10 = pain as bad as you can imagine.
  The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your worst pain during the last 24 hours prior to the visit".
Time Frame: Enrollment Visit (Day -14); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 445
units on a scale
  Enrollment Visit (N=438) | 7.6 (1.32)
  Baseline Visit (N=440) | 8.5 (1.11)
  Randomization Visit (N=377) | 5.8 (1.98)

9. Secondary Outcome: Open-label Titration Period: Comparative Double-blind Period Population Worst Mean Pain Intensity Scores Over the Past 24 Hours
Description: The recalled worst pain intensity during the last 24 hours was assessed using an 11-point Numeric Rating Scale (NRS), where 0 = "no pain" and 10 = "pain as bad as you can imagine".
  The participant was asked : "Please rate your pain intensity by assessing the one number that best describes your worst pain during the past 24 hours prior to the visit".
Time Frame: Enrollment Visit (Day-12); Baseline Visit (day 1); Randomization Visit (Day 22)
Population: Double-blind comparative population. Per Protocol Set (PPS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 7.8 (1.21) | 7.5 (1.27)
  Baseline Visit (N=139; N=149) | 8.5 (1.07) | 8.7 (0.97)
  Randomization Visit (N=139; N=149) | 6.3 (1.52) | 6.4 (1.4)

10. Secondary Outcome: Double-blind Comparative Period: Change in Worst Pain Intensity Over the Past 24 Hours
Description: The recalled worst pain intensity during the last 24 hours was assessed using an 11-point Numeric rating scale, where 0 = no pain and 10 = pain as bad as you can imagine.
  The participant was asked: "Please rate your pain intensity by assessing the one number that best describes your worst pain during the last 24 hours prior to the visit".
  A negative change indicates that the pain intensity decreased from the start of the trial.
Time Frame: Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-blind comparative population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale | -1.7 (2.67) | -1.8 (2.58)

11. Secondary Outcome: Open-label Titration Period: painDETECT Assessments
Description: The painDETECT was a participant completed questionnaire. The questionnaire consists of 14 questions in four domains. Based on these questions a final assessment score was calculated. The minimum score ranged from zero to a maximum of 38. Participants with a score between 0 and 12 were scored as being "negative" (had no neuropathic pain component). A value between 19 and 38 was rated as being "positive" (neuropathic component present). Values from 13 to 18 were scored as being "unclear".
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 445
units on a scale
  Enrollment Visit (N=438) | 21.4 (5.46)
  Baseline Visit (N=440) | 22.7 (5.74)
  Randomization Visit (N=377) | 16.9 (6.57)

12. Secondary Outcome: Open-label Titration Period: Comparative Double-blind Period Population painDETECT Assessment
Description: as for outcome 11
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-blind comparative population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 21.6 (5.23) | 21.7 (5.17)
  Baseline Visit (N=139; N=149) | 22.4 (5.21) | 23.8 (5.51)
  Randomization Visit (N=138; N=149) | 17.6 (5.93) | 18.4 (5.90)

13. Secondary Outcome: Double-blind Comparative Period: Change in painDETECT Final Assessment
Description: The painDETECT was a participant completed questionnaire. The questionnaire consists of 14 questions in four domains. Based on these questions a final assessment score was calculated. The minimum score ranged from zero to a maximum of 38. Participants with a score between 0 and 12 were scored as being "negative" (had no neuropathic pain component). A value between 19 and 38 was rated as being "positive" (neuropathic component present). Values from 13 to 18 were scored as being "unclear". The theoretical range of change in this trial ranged from -38 to 19. A negative change indicated a decrease in their neuropathic component of pain.
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-blind comparative population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 109 | 127
units on a scale
  Change from Baseline | -10.2 (8.57) | -11.0 (7.73)
  Change from Randomization | -6.0 (8.99) | -5.9 (7.22)

14. Secondary Outcome: Open-label Titration Period: Neuropathic Pain Symptom Inventory (NPSI) Overall Score Assessment
Description: In the Neuropathic Pain Symptom Inventory (NPSI) the participant rated their symptoms of neuropathic pain. Ten pain questions were answered on an 11-point scale; from 0 (symptom not present) to 10 (symptom at its worst imaginable intensity, e.g. worst burning imaginable). The overall NPSI score was calculated by the summation of all ten responses and ranges between 0 and 100. For pain descriptions burning, pressing, paroxysmal (pain like electric shocks or stabbing), evoked (due to touch) and paresthesia (sensation that is not unpleasant) or dysesthesia (unpleasant) sub-scores are reported. The overall values reported for all participants that completed the questionnaire are shown. A symptom was absent if the value is 0, the symptom was present in all participants and all participants rated it at its worst possible intensity if a value is 100.
Time Frame: Enrollment Visit; Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 445
units on a scale
  Overall Score Enrollment Visit (N=438) | 55.2 (16.86)
  Overall Score Baseline Visit (N=440) | 62.7 (18.41)
  Overall Score Randomization Visit (N=377) | 42.0 (20.29)

15. Secondary Outcome: Open-label Titration Period: Neuropathic Pain Symptom Inventory (NPSI) Overall Score Assessment in the Double-blind Comparative Period Population
Description: as for outcome 14
Time Frame: Enrollment Visit; Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-blind comparative population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Overall Score Enrollment Visit (N=138, N=149) | 54.8 (15.12) | 57.6 (16.07)
  Overall Score Baseline Visit (N=139, N=149) | 62.8 (17.13) | 65.4 (18.29)
  Overall Score Randomization Visit (N=139, N=149) | 45.2 (17.99) | 46.5 (18.57)
  Overall Score Final Evaluation Visit(N=131, N=143) | 28.9 (21.78) | 30.5 (22.38)

16. Secondary Outcome: Double-blind Comparative Period: Change in Neuropathic Pain Symptom Inventory (NPSI) Sub-scores and Overall Score Assessment
Description: In the Neuropathic Pain Symptom Inventory (NPSI) the participant rated their symptoms of neuropathic pain. Ten pain questions were answered on an 11-point scale, from 0 (symptom not present) to 10 (symptom at its worst imaginable intensity, e.g. Spontaneous Pressing Pain Subscore). The overall NPSI score was calculated by the summation of all ten responses and ranges between 0 and 100. For pain descriptions burning, pressing, paroxysmal (pain like electric shocks or stabbing), evoked (due to touch) and paresthesia (sensation that is not unpleasant) or dysesthesia (unpleasant) subscores are reported. The overall values reported for all participants that completed the questionnaire are shown. A symptom was absent if the value is 0, the symptom was present in all participants and all participants rated it at its worst possible intensity if a value is 10 (100 for the overall score) . A negative change indicates that the intensity of the symptom has decreased since the start of treatment.
Time Frame: Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-blind comparative population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 131 | 143
units on a scale
  Overall Score | -16.8 (18.95) | -16.6 (20.04)
  Subscore: Superficial Spontaneous Burning | -1.9 (2.75) | -2.3 (2.65)
  Subscore: Deep Sponatenous Pressing Pain | -1.4 (2.26) | -1.4 (2.58)
  Subscore: Paroxysmal Pain | -2.0 (2.39) | -1.6 (2.44)
  Subscore: Evoked Pain | -1.8 (2.28) | -1.7 (2.32)
  Subscore: Parasthesia/Dysesthesia | -1.4 (2.44) | -1.5 (2.49)

17. Secondary Outcome: Open-label Titration Period: Comparative Double-blind Period Population Short Form Health Survey (SF-12) Physical Health Composite Score (PCS)
Description: The Short Form Health Survey (SF-12) has several brief broad questions on 8 aspects of health (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. The physical and mental summary scores were calculated from the individual responses. A higher score indicates a better perceived state of health. All domains were scored on a scale from 0 (lowest level of health) to 100 (highest level of health), with 100 representing the best possible health state.
Time Frame: Enrollment Visit; Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 29.9 (8.55) | 29.8 (7.56)
  Baseline Visit (N=139; N=149) | 28.2 (8.17) | 28.5 (7.68)
  Randomization Visit (N=139; N=149) | 34.1 (9.36) | 34.1 (8.45)

18. Secondary Outcome: Double-blind Comparative Period: Changes in the Short Form Health Survey (SF-12) Physical Health Composite Score (PCS)
Description: The Short Form Health Survey (SF-12) has several brief broad questions on 8 aspects of health (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. The physical summary scores were calculated from the individual responses to those questions covering physical health. A higher score indicates a better participant perceived state of health. All domains were scored on a scale from 0 (lowest level of health) to 100 (highest level of health), with 100 representing the best possible health state.
  The change in the SF-12 score shows an improvement in health from baseline if the values are positive. The higher the value the greater the improvement.
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 131 | 143
units on a scale
  Change from Baseline Visit | 12.3 (12.98) | 11.1 (11.36)
  Change from Randomization Visit | 6.2 (13.04) | 5.6 (10.88)

19. Secondary Outcome: Open-label Titration Period: Comparative Double-blind Period Population Short Form Health Survey (SF-12) Mental Health Composite Score (MCS)
Description: The Short Form Health Survey (SF-12) has several brief broad questions on 8 aspects of health (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health) that a participant was asked to score over the last week. The mental health summary scores were calculated from the individual responses to two of the 12 questions. A higher score indicates a better participant perceived state of health. All domains were scored on a scale from 0 (lowest level of health) to 100 (highest level of health), with 100 representing the best possible mental health.
Time Frame: Enrollment Visit; Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 46.1 (11.84) | 44.8 (12.24)
  Baseline Visit (N=139; N=149) | 45.4 (12.43) | 43.2 (13.32)
  Randomization Visit (N=139; N=149) | 49.2 (11.64) | 47.3 (11.80)

20. Secondary Outcome: Double-blind Comparative Period: Change in Short Form Health Survey (SF-12) Mental Health Composite Score (MCS)
Description: as for outcome 19
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 131 | 143
units on a scale
  Change from Baseline Visit (N=131; N=143) | 3.9 (10.59) | 6.5 (11.62)
  Change from Randomization Visit (N=131; N=143) | 0.1 (8.42) | 2.5 (9.77)

21. Secondary Outcome: Open-label Titration Period: EuroQol-5 Dimension (EQ-5D) Health Status Index Score for the Double-blind Comparative Period Population
Description: The participant scored the EuroQol-5 questionnaire. The EuroQol-5 questionnaire uses a health state classification with 5 dimensions. Each dimension was assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1 (with 1 indicating "full health" and 0 representing "dead"). The higher the values (the closer the value is to 1) the better the health status in a treatment group.
Time Frame: Enrollment Visit (day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 0.32 (0.304) | 0.33 (0.313)
  Baseline Visit (N=139; N=149) | 0.29 (0.306) | 0.18 (0.316)
  Randomization Visit (N=139; N=149) | 0.55 (0.254) | 0.52 (0.237)

22. Secondary Outcome: Double-blind Comparative Period: Change EuroQol-5 Dimension (EQ-5D) Health Status Index
Description: as for outcome 21
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 131 | 143
units on a scale
  Change from Baseline Visit | 0.34 (0.358) | 0.43 (0.386)
  Change from Randomization Visit | 0.09 (0.317) | 0.09 (0.254)

23. Secondary Outcome: Double-blind Comparative Period: Patient Global Impression of Change (PGIC)
Description: In the Patient Global Impression of Change (PGIC) the participant indicated the perceived change over the treatment period. PGIC is a 7 point scale where the patient's rates overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Time Frame: Randomization Visit (Day 22) to Final Evaluation Visit (Day 77)
Population: Double-blind comparative population. Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 152 | 157
participants
  Very much improved | 28 | 32
  Much improved | 44 | 66
  Minimally improved | 51 | 31
  No change | 10 | 10
  Minimally worse | 5 | 5
  Much worse | 4 | 5
  Very much worse | 0 | 1
  Missing | 10 | 7

24. Secondary Outcome: Double-blind Comparative Period: Clinician Global Impression of Change (CGIC)
Description: In the Clinician Global Impression of Change (CGIC) the clinician indicated the perceived change over the treatment period. The clinician was requested to choose one of seven categories for each participant. The Clinician rated the participants change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Time Frame: Randomization Visit (Day 22) to Final Evaluation Visit (Day 77)
Population: Double-Blind Comparative Population. Full Analysis Set (FAS).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 142 | 150
participants
  Very much improved | 26 | 30
  Much improved | 54 | 82
  Minimally improved | 46 | 19
  No change | 8 | 10
  Minimally worse | 3 | 2
  Much worse | 5 | 5
  Very much worse | 0 | 2
  Missing | 10 | 7

25. Secondary Outcome: Open-label Titration Period: Hospital Anxiety and Depression Scale - Anxiety in the Double-blind Comparative Period Population
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe anxiety. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate anxiety. A score of 11 or above is considered to be a case of anxiety.
  A decrease in values over the trial period indicate that there has been an improvement.
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 7.4 (4.51) | 8.6 (4.94)
  Baseline Visit (N=139; N=149) | 7.7 (4.52) | 9.0 (5.15)
  Randomization Visit (N=139; N=149) | 5.8 (3.77) | 7.1 (4.39)

26. Secondary Outcome: Double-blind Comparative Period: Change in Hospital Anxiety and Depression Scale - Anxiety in the Double-blind Comparative Period Population
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe anxiety. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate anxiety. A score of 11 or above is considered to be a case of anxiety.
  A negative sign indicates that there has been a decrease in anxiety since the start of treatment.
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 123 | 137
units on a scale
  Change from Baseline Visit | -2.2 (3.70) | -3.1 (4.28)
  Change from Randomization Visit | -0.3 (2.93) | -1.2 (3.38)

27. Secondary Outcome: Open-label Titration Period: Hospital Anxiety and Depression Scale - Depression in the Double-blind Comparative Period Population
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe depression. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate depression. A score of 11 or above is considered to be a case of depression. A decrease in values over time indicates that there has been an improvement.
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-blind Comparative Population; Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
units on a scale
  Enrollment Visit (N=138; N=149) | 6.9 (4.18) | 7.8 (4.43)
  Baseline Visit (N=139; N=149) | 7.6 (4.66) | 8.6 (4.81)
  Randomization Visit (N=139; N=149) | 6.0 (3.96) | 6.8 (4.24)

28. Secondary Outcome: Double-blind Comparative Period: Change in Hospital Anxiety and Depression Scale - Depression in the Double-blind Comparative Period Population
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-assessment scale for the symptom severity of anxiety disorders and depression. It comprises 14 items. Seven statements describe depression. Each answer is scored on a four-point scale (0-3). All seven answers are summed to a total score with a maximum score of 21 points. A score below 7 is not considered to indicate depression. A score of 11 or above is considered to be a case of depression. A decrease in values over time indicates that there has been an improvement. A negative change value indicates a decrease in the depression score since the start of treatment.
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22); Final Evaluation Visit (Day 77)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 123 | 137
units on a scale
  Change from Baseline Visit | -2.0 (3.56) | -3.1 (3.99)
  Change from Randomization Visit | -0.4 (3.06) | -1.3 (2.94)

29. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Latency
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the sleep latency.
  To assess latency the participant was asked: How long after bedtime/lights out did you fall asleep last night [hours]?
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Enrollment Visit (Day -12): Participant feedback at the Enrollment Visit; on previous analgesic medication prior to study drug start.
- Baseline Visit (Day 1): At the end of the washout period prior to starting 100 mg/day tapentadol prolonged release.
- Randomization Visit (Day 22): End of open-label titration period. Participants with 100 to 300 mg/day tapentadol.
Arm/Group | Enrollment Visit (Day -12) | Baseline Visit (Day 1) | Randomization Visit (Day 22)
Number analyzed (Participants) | 438 | 440 | 377
hours | 1.2 (1.50) | 1.5 (1.56) | 1.3 (1.67)

30. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Latency in the Double-blind Comparative Period Population
Description: The sleep evaluation questionnaire was completed by the participant. The participant was asked: How long after bedtime/lights out did you fall asleep last night [hours]? The values are for the night prior to the Randomization Visit (Baseline) and for the night prior to the Final Evaluation Visit (12 weeks after randomization). The higher the value the longer it took to fall asleep. Sleep evaluation questionnaire (SQ) items
Time Frame: Enrollment Visit (Day -12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
hours
  Enrollment Visit (N=138, N=149) | 1.3 (1.70) | 1.3 (1.52)
  Baseline Visit (N=139, N=149) | 1.5 (1.65) | 1.5 (1.54)
  Randomization Visit (N=139, N=149) | 1.1 (1.45) | 1.4 (1.78)

31. Secondary Outcome: Double-blind Comparative Period Sleep Evaluation Questionnaire: Change in Latency
Description: The sleep evaluation questionnaire was completed by the participant. The participant was asked: How long after bedtime/lights out did you fall asleep last night [hours]? The values are for the night prior to the visits. The negative change from baseline indicates that the time to falling asleep decreased from baseline in a treatment group.
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22) to Final Evaluation Visit (Day 77)
Population: Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 123 | 137
hours
  Change from baseline visit | -0.3 (2.30) | -0.3 (2.10)
  Change from randomization visit | 0.2 (1.88) | -0.2 (2.04)

32. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Number of Awakenings
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the number of awakenings.
  How many times did you wake up during the night? The values were calculated from the data that participants self-reported for the night prior to their Randomization Visit (Baseline), for the night prior to the Baseline Visit (Day 1) and the night prior to the Randomization Visit (Day 22).
  The participant was asked at each visit: "How many times did you wake up during the night?"
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | Enrollment Visit (Day -12) | Baseline Visit (Day 1) | Randomization Visit (Day 22)
Number analyzed (Participants) | 438 | 440 | 377
Number of Awakenings | 3.3 (2.64) | 3.9 (3.11) | 2.5 (1.87)

33. Secondary Outcome: Open-label Titration Period: Sleep Evaluation - Number of Awakenings in the Double-blind Comparative Period Population
Description: as for outcome 32
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
Number of Awakenings
  Enrollment Visit (N=138; N=149) | 3.2 (2.84) | 3.4 (2.36)
  Baseline Visit (N=139; N=149) | 3.6 (2.47) | 4.6 (4.01)
  Randomization Visit (N=139; N=149) | 2.5 (1.76) | 2.7 (2.00)

34. Secondary Outcome: Double-blind Comparative Period: Change in the Number of Awakenings
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the number of awakenings. Participants were asked: How many times did you wake up during the night? The change in the Number of Awakenings was calculated from the data that participants self-reported for the night prior to their Randomization Visit (Baseline), for the night prior to the Baseline Visit (Day 1) and the night prior to the Final Evaluation Visit (Day 77). A negative change indicates that the number of awakenings in a treatment group have gone down since the Baseline or Randomization Visit. In general pain can interfere with sleep, one potential indicator is the number of awakenings.
Time Frame: Baseline Visit (Day 1); Randomization Visit (Day 22) to Final Evaluation Visit (Day 77)
Population: Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 123 | 137
Number of Awakenings
  Change from Baseline Visit | -1.4 (2.57) | -2.5 (3.11)
  Change from Randomization Visit | -0.2 (2.01) | -0.8 (1.78)

35. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Time Slept
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the number of awakenings.
  The participant was asked: "How long did you sleep last night?" [Answered in hours and minutes].
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enrollment Visit (Day -12) | Baseline Visit (Day 1) | Randomization Visit (Day 22)
Number analyzed (Participants) | 438 | 440 | 377
hours | 5.8 (1.69) | 5.3 (1.79) | 6.4 (1.41)

36. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Number of Hours Slept in the Double-blind Comparative Period Population
Description: The participants were requested to answer the following question:
  How long did you sleep last night [hours]? The values were calculated from the data that participants self-reported for the night prior to their Randomization Visit (Baseline) and for the night prior to the End of the Continuation Visit (12 weeks after randomization).
Time Frame: Enrollment Visit (Day -12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Per Protocol Set (PPS).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
hours
  Enrollment Visit (N=138, N=149) | 5.8 (1.66) | 5.7 (1.70)
  Baseline Visit (N=139, N=149) | 5.3 (1.67) | 5.2 (1.70)
  Randomization Visit (N=139, N=149) | 6.2 (1.30) | 6.4 (1.59)

37. Secondary Outcome: Double-blind Comparative Period: Sleep Evaluation Questionnaire - Change in the Number of Hours Slept
Description: The sleep evaluation questionnaire was completed by the participant. The answer was in response to the question: Sleep evaluation: How long did you sleep last night [hours]? The value reported is the change in the number of hours of sleep from baseline. The positive value indicates that there was an increase in the number of hours of sleep in a treatment group.
Time Frame: Baseline Visit (Day -12); Randomization Visit (Day 1); Final Evaluation Visit (Day 77)
Population: Per Protocol Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 123 | 137
hours
  Change from baseline visit | 1.2 (1.89) | 1.6 (1.84)
  Change from randomization visit | 0.3 (1.71) | 0.3 (1.70)

38. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Overall Quality of Sleep
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the overall quality of sleep.
  The participant rated this categorically as being one of the following: excellent, good, fair or poor.
Time Frame: Enrollment Visit (Day-12); Baseline Visit (Day 1); Randomization Visit (Day 22)
Population: Observed.
Measure: Number; unit: participants
Arm/Group | Enrollment Visit (Day -12) | Baseline Visit (Day 1) | Randomization Visit (Day 22)
Number analyzed (Participants) | 445 | 445 | 445
participants
  Excellent | 9 | 5 | 21
  Good | 110 | 76 | 173
  Fair | 171 | 149 | 127
  Poor | 148 | 210 | 56
  Missing | 7 | 5 | 68

39. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Overall Quality of Sleep in the Double-blind Comparative Period Population
Description: as for outcome 38
Time Frame: Enrollment Visit (Day-12)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
participants
  Excellent | 1 | 5
  Good | 37 | 30
  Fair | 42 | 61
  Poor | 58 | 53
  Missing | 1 | 0

40. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Overall Quality of Sleep in the Double-blind Comparative Period Population
Description: as for outcome 38
Time Frame: Baseline Visit (Day 1)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
participants
  Excellent | 2 | 1
  Good | 23 | 17
  Fair | 42 | 49
  Poor | 72 | 82

41. Secondary Outcome: Open-label Titration Period: Sleep Evaluation Questionnaire - Overall Quality of Sleep in the Double-blind Comparative Period Population
Description: as for outcome 38
Time Frame: Randomization Visit (Day 22)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
participants
  Excellent | 7 | 8
  Good | 62 | 59
  Fair | 48 | 56
  Poor | 22 | 26

42. Secondary Outcome: Double-blind Comparative Period: Change in the Overall Quality of Sleep
Description: The sleep evaluation questionnaire was completed by the participant. The questionnaire measures 4 main concepts: 1 of the 4 main concepts being the overall quality of sleep.
  The improvement, no change or worsening is reported based on the replies scored by the participants given at their End of Continuation Visit.
Time Frame: Randomization Visit (Day 22) to Final Evaluation (Day 77)
Population: Double-Blind Comparative Population. Per Protocol Set (PPS).
Measure: Number; unit: participants
Arm/Group | Tapentadol Prolonged Release | Tapentadol Prolonged Release and Pregabalin
Number analyzed (Participants) | 139 | 149
participants
  Improvement | 39 | 58
  No change | 63 | 59
  Worsening | 21 | 20
  Missing | 16 | 12

43. Secondary Outcome: Open-label Titration Period: Subject's Satisfaction With Treatment
Description: Participants rated their satisfaction with the study drug (IMPs) by answering the following question on a 5-point rating scale:
  "How would you rate your overall satisfaction with your current pain treatment?": Excellent, Very Good, Good, Fair and Poor.
Time Frame: End of Open-label Titration Period at Randomization Visit (Day 22)
Population: Last Observation Carried Forward (LOCF); Per Protocol Set
Measure: Number; unit: participants
Groups:
- Tapentadol Prolonged Release: Tapentadol PR (100 - 300 mg per day) oral administration twice daily in the open-label titration period.
Arm/Group | Tapentadol Prolonged Release
Number analyzed (Participants) | 445
participants
  Poor | 12
  Fair | 119
  Good | 178
  Very Good | 58
  Excellent | 11
  Missing | 67

44. Secondary Outcome: Double-blind Comparative Period: Subject's Satisfaction With Treatment
Description: as for outcome 43
Time Frame: End of Comparative Period at Final Evaluation Visit (Day 77)
Population: Last Observation Carried Forward (LOCF); Per Protocol Set
Measure: Number; unit: participants
Groups:
- Tapentadol in the Comparative Period: The dose of Tapentadol Prolonged Release was increased to 400 mg (2 x 200mg) and a week later to 500 mg (2 x 250 mg) per day and maintained at 500 mg per day.
- Tapentadol and Pregabalin in the Comparative Period: Tapentadol Prolonged Release 300 mg per day (2 x 150 mg) plus Pregabalin 2 x 75 mg (total daily dose of 150 mg). A week later the dose of Pregabalin was increased to a total daily dose of 300 mg per day (2 x 150 mg), the Tapentadol Prolonged Release dose remained at 300 mg per day.
Arm/Group | Tapentadol in the Comparative Period | Tapentadol and Pregabalin in the Comparative Period
Number analyzed (Participants) | 139 | 149
participants
  Poor | 3 | 6
  Fair | 32 | 28
  Good | 43 | 43
  Very Good | 32 | 43
  Excellent | 21 | 23
  Missing | 8 | 6

ADVERSE EVENTS:
Time Frame: Baseline Visit; up to end of Week 11.
Description: Treatment Emergent Adverse Events are reported, starting with the first dose in the open-label titration period on Day 1 up to Day 77. TEAEs are reported up to Day 91 at the End of the Follow-Up visit.
  One participant died, before the baseline visit, during the washout phase of the clinical trial.
Groups:
- Open-Label Tapentadol Titration Period: During the 3-week Titration Period, Tapentadol Prolonged Release was administered in an open-label fashion.
  Titration dose steps on a weekly basis:
  First 50 mg administered twice daily, then 100 mg administered twice daily and then 150 mg administered twice daily.
  The titration period could be shortened to 10 days, with a participant at a predefined dose level for at least 3 days.
  The dose of 300 mg Tapentadol per day was maintained until the Randomization Visit.
- Open-Label Tapentadol Pick-Up Arm: Participants that drop-out of the Comparative Period, due to tolerability issues, were permitted to continue on Tapentadol Prolonged Release at either 300 mg per day or 400 mg per day.
- Open-Label Tapentadol Continuation Period: Participants who did not qualify for randomization to the Comparator Period, continued on a stable dose of Tapentadol Prolonged Release 300 mg per day if they had reached a satisfactory level of pain relief.
Arm/Group | Open-Label Tapentadol Titration Period | Tapentadol in the Comparative Period | Tapentadol and Pregabalin in the Comparative Period | Open-Label Tapentadol Pick-Up Arm | Open-Label Tapentadol Continuation Period
Serious Adverse Events (participants affected / at risk) | 3/445 | 5/154 | 3/159 | 2/37 | 2/59
Other Adverse Events (participants affected / at risk) | 227/445 | 98/154 | 103/159 | 37/37 | 36/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Tapentadol Titration Period (N=445) | Tapentadol in the Comparative Period (N=154) | Tapentadol and Pregabalin in the Comparative Period (N=159) | Open-Label Tapentadol Pick-Up Arm (N=37) | Open-Label Tapentadol Continuation Period (N=59)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 0 | 0 | 0 | 0 — Luxation of new implanted total endoprosthesis left hip
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Tapentadol Titration Period (N=445) | Tapentadol in the Comparative Period (N=154) | Tapentadol and Pregabalin in the Comparative Period (N=159) | Open-Label Tapentadol Pick-Up Arm (N=37) | Open-Label Tapentadol Continuation Period (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Brachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular Disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Palpitation (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Cupulolithiasis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Ear Discomfort (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
External Ear Disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Inner Ear Disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Motion Sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 0
Accommodation Disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 1 | 0 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pruritis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 2 | 0 | 3 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual Impairment (Eye disorders) | 0 | 1 | 2 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 2 | 2 | 1 | 1
Abdominal Symptom (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abnormal Faeces (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colonic Polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 25 | 11 | 8 | 9 | 10
Diarrhoea (Gastrointestinal disorders) | 14 | 6 | 3 | 3 | 2
Dry Mouth (Gastrointestinal disorders) | 35 | 6 | 8 | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 6 | 1 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Flatuence (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 58 | 16 | 14 | 12 | 11
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Uvulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 20 | 9 | 5 | 5 | 4
Asthenia (General disorders) | 6 | 4 | 0 | 2 | 2
Chest Discomfort (General disorders) | 2 | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 1 | 0 | 1 | 0
Drug Withdrawal Syndrome (General disorders) | 2 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 25 | 13 | 16 | 10 | 5
Feeling Abnormal (General disorders) | 2 | 0 | 1 | 0 | 0
Feeling Cold (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling Drunk (General disorders) | 1 | 1 | 2 | 1 | 0
Feeling Hot (General disorders) | 1 | 0 | 0 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 2 | 0 | 0
Generalised Oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Hyperplasia (General disorders) | 0 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Influenza Like Illness (General disorders) | 4 | 2 | 3 | 1 | 0
Irritability (General disorders) | 3 | 0 | 3 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 1 | 0
Oedema Peripheral (General disorders) | 6 | 0 | 3 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acute Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes Zoster Oticus (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 2 | 5 | 2 | 3
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis Media Acute (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 1 | 1 | 2
Vaginal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Creatinine Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 2 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Lasegue's Test Positive (Investigations) | 0 | 0 | 1 | 0 | 1
Lipase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neurological Examination Abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Nitrite Urine Present (Investigations) | 1 | 0 | 0 | 0 | 0
Prostatic Specifc Antigen Increased (Investigations) | 0 | 0 | 2 | 0 | 0
Protein Urine Present (Investigations) | 0 | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 3 | 0 | 0 | 1
White Blood Cell Count Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 12 | 2 | 1 | 3 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Intervertebral Disc Protusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 3 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 0 | 1
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Allodynia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 2 | 2 | 2 | 3 | 0
Carotid Arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 51 | 17 | 28 | 11 | 9
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 3 | 0 | 0
Dyskinesia (Nervous system disorders) | 3 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 40 | 10 | 13 | 5 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 1 | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 2 | 1 | 2 | 0 | 0
Mental Impairment (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Movement Disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Muscle Contraction Involuntary (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 5 | 1 | 0 | 2 | 0
Restless Leg Syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sensory Loss (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 29 | 13 | 19 | 11 | 4
Speech Disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tension Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 3 | 2 | 2 | 0 | 2
Abnormal Dreams (Psychiatric disorders) | 3 | 0 | 2 | 1 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 4 | 3 | 3 | 1
Apathy (Psychiatric disorders) | 2 | 0 | 0 | 0 | 2
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depressed Mood (Psychiatric disorders) | 4 | 3 | 3 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Drug Dependence (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Emotional Disorder (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Fear (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Food Aversion (Psychiatric disorders) | 1 | 1 | 0 | 2 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Initial Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 3 | 5 | 3 | 3
Libido decreased (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Listless (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
Middle Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mood Swings (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Mood Altered (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 1 | 2 | 1 | 2
Nightmare (Psychiatric disorders) | 1 | 0 | 1 | 0 | 3
Restlessness (Psychiatric disorders) | 5 | 1 | 1 | 1 | 2
Sleep Disorder Due To General Medical Condition, Insomnia Type (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Sleep Talking (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 4 | 2 | 2 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Tic (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Bladder Discomfort (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 3 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0
Micturition Disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal Cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast Swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 2 | 1 | 0
Sexual Dysfunctio (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 1 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 21 | 18 | 10 | 10 | 5
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 6 | 1 | 4 | 2
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin Tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Blood Pressure Fluctuation (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Flushing (Vascular disorders) | 2 | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 10 | 0 | 0 | 3 | 1
Hypertension (Vascular disorders) | 3 | 1 | 5 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.